CLINICAL TRIAL: NCT02715661
Title: Cerebrovascular Outcomes in Ischemic Heart Disease Patients Undergoing Cardiac Rehabilitation
Brief Title: Cerebrovascular Outcomes in Ischemic Heart Disease
Acronym: IHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Kevin Shoemaker, Dr. Kevin Shoemaker, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 107620
Record Dates: First submitted 2016-03-07; First posted 2016-03-22 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Cardiovascular Disease
Keywords: blood flow; brain health; exercise; endothelial activation
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Coronary artery disease (Active Comparator): those with a diagnosis of coronary artery disease having been hospitalized for a cardiac event. The intervention is six-month interval of exercise .
  Interventions: Other: exercise
- Metabolic Syndrome (Active Comparator): Metabolic Syndrome patients are defined by having Systolic Blood Pressure (SBP)>130 and/or Diastolic Blood Pressure (DBP)>85 mmHg and any two of the following criteria: Abdominal obesity (waist circumference >102cm in males;>88cm in females), Fasting triglycerides > 1.695 mmol/L, Low HDL cholesterol: Males < 1.04 mmol/L; Females < 1.29 mmol/L, Fasting glucose >5.60 mmol/L. Participants will be assigned randomly into an exercise and a delayed exercise intervention, 6 months.
  Interventions: Other: exercise
- Health Control (Active Comparator): Control individuals will have no diagnosis of cardiac, vascular, metabolic, inflammatory or neurological disease, and have not been on any medication for such conditions in the past 12 months. Participants will be assigned randomly into an exercise and a delayed exercise intervention, 6 months.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — six-month interval of exercise

SUMMARY:
This project will examine the association between (cardio)vascular disease, blood supply to the brain, and cerebrovascular endothelial activation. Also, we will investigate the impact of exercise rehabilitation on brain vascularization, cerebrovascular endothelial function and blood flow control.

DETAILED DESCRIPTION:
This is a randomized control trial, with randomization nested within rationally-formed groups. Three major groups will be assessed: 1) Coronary artery disease (CAD) patients, 2) Metabolic Syndrome (MetS), and 3) healthy Control (CTL) participants. Allocation into the Healthy CTL versus MeTS groups will be confirmed at the pre-study screening visit based on medical questionnaires, blood sample outcomes, and ultrasound imaging (see below). All CTL and MeTS participants will be allocated by random assignment to a six-month exercise training group, or a 6-month "wait-list" training group followed by a 6-month exercise training period. The exercise training will be in accordance with American College of Sports Medicine and Canadian Society for Exercise Physiology guidelines supporting 3 days/week in the laboratory with target heart rate-based aerobic activity (~30 minutes/day) and two days of at-home activity. Based on target heart rate, levels of exercise intensity and/or duration will be adjusted every two weeks to sustain the training stimulus. CAD patients are defined here as those with a diagnosis of coronary artery disease having been hospitalized for a cardiac event. Within the recruited CAD participants, Group 1 (CADcr) will volunteer to receive a structured cardiac rehabilitation (CR) program. Group 2 (CADuc) will receive the recommendation for cardiac rehabilitation and choose not to participate (due to various reasons including distance to cardiac rehabilitation site), yet volunteer to the testing procedures at baseline and following a six month period. While random assignment is preferred, it is not feasible in CAD patients because, in our experience, geographical constraints or other personal barriers restrict access to CR and because CR is often considered the normal standard of care (they won't volunteer to avoid CR if they want CR). Instead, a naturalistic control approach will be used whereby patients who do not participate in CR may still participate by undergoing the testing before and following a six month period of time. Use of recall surveys will establish activity patterns in the non-exercise training groups or wait periods. Both groups will receive the same in-hospital education, referral to a CR program, personal prescription (referral), encouragement and follow-up. All subjects will complete a series of tests before and following the six-month interval of exercise or time control. Exercise training and the majority of testing will occur in the Laboratory for Brain and Heart Health (Labatt Health Sciences Building, Rm 402). Protocols: Cardio-respiratory Fitness: Fitness will be determined using a self-paced six-minute walk test (6MWT) that will be administered as per American Thoracic Society (ATS) guidelines whereby a physician's presence is not required. Blood Sample: After resting quietly for up to 30 min, a fasting (>3 hours) venous blood sample will be taken from the antecubital vein for analysis of blood glucose, lipids, and insulin (LifeLabs), markers of astrocyte and vascular damage (D. Fraser), endothelial function (e.g. endothelin, P-selectin) and inflammation (e.g. hsCRP, TNFa, IL-1, IL-6, IL-10), neural function markers (e.g. epinephrine, norepinephrine), and proliferative factors (e.g. NFK-B, brain-derived neurotrophic factor (BDNF), VEGF) (K. Summers). Additional samples of 10 mL whole blood will be taken to Robarts Research Institute for analysis of genetic markers of vascular risk (e.g. Apolipoprotein E (APOE) or BDNF polymorphisms (R. Hegele)) and for monocyte inflammatory profiles using flow-cytometry (G. Dekaban). Up to 5 samples of plasma (~1 mL) will be sent to Victoria Hospital for cell culture fluid-flow analysis of polymorphonuclear cell binding (G. Cepinskas). The total volume of blood sample will not exceed 60 mL. Vascular Ultrasound: Ultrasound will be used to measure artery diameters and blood flow in the Carotid Artery, Carotid Sinus, Brachial Artery and Femoral Artery. Dilation of the brachial artery will also be measured following five minutes of forearm ischemia (flow-mediated dilation) and for four minutes following a sublingual single dose (0.4 mg) of sodium nitroglycerine (standard over-the-counter self-treatment for angina). Sympathetic Nerve Activity: Peripheral sympathetic nerve activity will be obtained from the peroneal nerve using microneurography. A 200 µm-diameter, 35 mm long tungsten microelectrode tapered to an uninsulated 1- to 5-µm tip is inserted transcutaneously into the peroneal nerve just posterior to the fibular head. A reference electrode is positioned subcutaneously 1-3 cm from the recording site. A sympathetic nerve site is confirmed by the characteristic pulse-synchronous burst pattern that does not produce skin paraesthesias and that increases in frequency during a voluntary apnea and/or a Valsalva manoeuvre but not during arousal to a loud noise. Transcranial Ultrasound: A small probe held against each of the temporal windows (just behind the eyes) with a headband will measure flow velocity within the middle and/or posterior cerebral arteries. Cerebrovascular Reactivity (Hypercapnia): Subjects will breathe a hypercapnic gas mixture of 5% CO2/21% O2/Balance N2 through a 2-way non-rebreathing valve. This gas will be inspired for up to 5 minutes in each of two repeated trials separated by at least 5 minutes of recovery. Sit-to-stand test: To test dynamic rate of recovery in cerebral blood flow during transient changes in blood pressure, brain blood flow by transcranial Doppler ultrasound, blood pressure, heart rate, and end tidal CO2 (with a mask) will be measured during ~3 min of seated rest, two minutes of standing, and then a period of seated rest. This protocol may be repeated up to three times. A gas analyzer and face mask mechanism will enable measurement of expired oxygen and carbon dioxide in each of the hypercapnia and sit-to-stand tests. Electrocardiogram: A standard electrocardiogram will be collected via small surface electrodes on the chest to determine heart rate. Ventilation Patterns: A respitrace strain gauge will be placed around the chest to record breathing patterns. Blood pressure will be measured using a small cuff place on a finger (Finometer), and confirmed with upper arm sphygmomanometry. Hemoglobin saturation will be measured by a pulse oximeter on one of the digits. 1. 6-min walk test: Using a self-paced format, participants will walk back and forth along a long hallway for six minutes while the distance covered will be recorded. Participants may rest as needed throughout the test. 2. Leg and arm muscle strength (isometric). Participants will push a single arm or leg against a resistance machine while the force is measured. Three maximal-effort 3-sec repetitions will be repeated separated by a minute or two of rest. Neuropsychology Tests: These tests will study the key functional outcomes in vascular cognitive impairment and include measures related to mood, memory and cognition. The tests are pen-and-paper, will be administered by trained personnel, and, based on published standards (Hachinski et al., 2006) will include the following: Overall Cognitive Function: Montreal Cognitive Assessment (MOCA), Trail making test, and The Stroop Word-Colour Test. The latter task takes advantage of our ability to read words more quickly and automatically than we can name colors. Executive Function (Animal Naming, Controlled Oral Word), Association (Trail Making Test); Language (Boston Naming Test 2nd Edition, short form); Visuospatial (Rey-Osterrieth Complex, Figure Copy, Complex Figure Memory); Digit Span and Digit Symbol coding from the Wechsler Adult Intelligence Scale IV (WAIS-III; with Canadian norms) Memory (Rey Auditory Verbal Learning Test; http://www.wpspublish.com/store/Search?Q=Rey%20Auditory%20Verbal%20Learning%20Test%E2%84%A2%20(RAVLT%E2%84%A2); NOTE: In an attempt to address the practice effect problem related to repeated trials of the same test, alternate forms of some scales may be administered in a counter-balanced manner when appropriate. (Reference: V. Hachinski et al. National Institute of Neurological Disorders and Stroke - Canadian Stroke Network Vascular Cognitive Impairment Harmonization Standards, Stroke, 2006, 37:2220-2241) Magnetic Resonance Imaging (MRI): Two separate MRI protocols will be performed by each participant. These will be completed on either the 3 Tesla or 7 Tesla imaging systems at Robarts. The series of images acquired will include: 1) T1 MPRAGE anatomical, 2) FLAIR for white matter hyperintensities, 3) MR angiography for vascular architecture, 4) black-blood angiography of middle cerebral artery at baseline and again after up to five minutes of hypercapnia. Sample Schedule of Testing: These will be performed at each of the pre and post training periods. Visit 1 - Laboratory Testing 1 (3 hours) Consent: 15 min Supine rest: 30 min Blood samples: 10 min (used partly for group allocation in the pre test) Snack: 10 min Instrumentation (including transcranial Doppler and carotid artery vascular ultrasound imaging): 60 min Cerebrovascular Reactivity to hypercapnia and sit-to-stand tasks: 45 min Visit 2 - Laboratory Testing 2 (2h) Cognitive tests: 45 min Vascular imaging: 30 min Six-min walk: 10 min Leg Muscle Strength: 10 min Visit 3 - MRI Testing (<1.5 hours total time) Baseline blood pressure: 10 min MRI Preparation: 10 min Anatomical: 10 min White Matter Hyperintensities: 10 min Angiography: 20 min MR angiography of middle cerebral artery with hypercapnia: 20 min The Interventions: Rehabilitative Exercise: The cardiac rehabilitation (CR) programs will provide the initial exercise intervention for referred CAD patients (Dr. Suskin). The CR program uses standardized, prescriptive and progressive exercise (primarily aerobic exercise) practices to improve the functional capacity of patients following a clinical cardiac intervention. The CR program in London lasts for 6 months. In general, aerobic exercise training is at an intensity of 40%-70% heart rate reserve or, a rate of perceived exercise score of 11-14 (on the 6-20 Borg scale), 3-7 d/wk, at 20-60 min/session (or multiple 10-min sessions).

ELIGIBILITY:
Inclusion Criteria:

Coronary Artery Disease

* inclusion age range is 45-80 years of age
* both female and male participants are being studied
* upon discharge from hospital, are referred into Cardiac Rehabilitation (CR) programs in London. Prospective able to read & write English
* living in private residence
* under the care of a family physician, having been discharged from hospital following admission for acute coronary syndrome (e.g. ST elevation or non ST elevation MI), angina, per cutaneous coronary intervention (PCI), or coronary artery bypass graft (CABG) as documented by the attending physician.
* Coronary artery disease patients who were not eligible for cardiac rehabilitation or who were referred to CR but have declined (by not enrolling or attending CR) will be invited as Usual Care (CADuc) Coronary artery disease Subjects.

Metabolic Syndrome Group:

* inclusion age range is 45-80 years of age
* both female and male participants are being studied
* Systolic Blood Pressure>130 and/or Diastolic Blood Pressure>85 mmHg
* any two of the following criteria:
* Abdominal obesity (waist circumference >102cm in males;>88cm in females), Fasting triglycerides > 1.695 mmol/L, Low HDL cholesterol: Males < 1.04 mmol/L; Females < 1.29 mmol/L, Fasting glucose >5.60 mmol/L
* able to read & write English
* living in private residence

Healthy Control Group

* the inclusion age range is 18-80 years of age
* both female and male participants are being studied
* Control individuals will have no diagnosis of cardiac, vascular, metabolic, inflammatory or neurological disease, and have not been on any medication for such conditions in the past 12 months able to read & write English
* living in private residence

Exclusion Criteria:

* As magnetic resonance imaging (MRI) is used to examine the brain in this study, participants will not be included in the study if they have any history of head or eye injury involving metal fragments, some type of implanted electrical device (such as a cardiac pacemaker). If they have severe heart disease (including susceptibility to heart rhythm abnormalities), they should not have an MRI scan unless supervised by a physician. Additionally they should not have a MRI scan if they have conductive implants or devices such as skin patches, body piercing or tattoos containing metallic inks because there is a risk of heating or induction of electrical currents within the metal element causing burns to adjacent tissue. In addition to these guidelines, patients with claustrophobia will not be studied in the MRI elements of this project.
* respiratory disease
* a history of psychosis
* eating disorders
* manic or bipolar disorder
* major psychiatric conditions
* immunological, congenital or neurodegenerative disorders (e.g., Raynaud's syndrome, multiple sclerosis, Parkinson's Disease, ALS),
* dependence on alcohol or drugs within the past year
* who smoke (within the past five years)
* women who are pregnant or trying to become pregnant will also be excluded
* participants will be excluded if they are unable to provide written informed consent, or to complete questionnaires or health history forms due to language or cognitive difficulties
* coronary artery disease Subjects will be excluded if they have:
* unstable heart rhythm
* congenital coronary abnormality
* cardiomyopathy
* severe congestive heart failure
* 2°-3° atrioventricular block
* more than 2 M.I.s
* major arrhythmias such as atrial fibrillation or more than 4 ectopic beats/min, sick sinus syndrome, or are scheduled to undergo PCI or CABG within 2 months following hospital discharge
* all healthy Control and Metabolic Syndrome participants will provide clearance from their Family Physician to participate in exercise training on the Physical Activity Readiness Questionnaire (PARQ) Form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-03; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
cerebrovascular properties | baseline and 6 months
  This will be measured first by the change in blood flow velocity through the middle cerebral artery in response to the 5% CO2/95% O2 challenge and a sit-to-stand manoeuvre. Measures will be made using transcranial Doppler. Subsequently, the diameter of the middle cerebral artery will be measured with MRI T2 sequences (time of flight) at 7Tesla.
  Multiple measurements will be aggregated to arrive at one reported value of cerebrovascular reactivity to carbon dioxide.

SECONDARY OUTCOMES:
1) vascular cognitive impairment | baseline and 6 months
  These will be made with pen-and paper questionnaires identified above.
2) Brain grey matter and white matter mass, white matter hyperintensities | baseline and 6 months
  This is measured from the MRI T1 anatomical and FLAIR sequences.
  Multiple measurements will be aggregated to scientifically examine the association between (cardio)vascular disease, blood supply to the brain, and cerebrovascular endothelial activation. These measurements will allow us to investigate the impact of exercise rehabilitation on brain vascularization, cerebrovascular endothelial function and blood flow control.
3) blood borne markers of inflammation | baseline and 6 months
  will be measured using multiplex and ELISA technology,
4) vascular endothelial damage | baseline and 6 months
  will be assessed using ultrasound imaging analysis of intima-media thickness (Carotid artery) and the flow-mediated dilation of the brachial artery.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Shoemaker, PhD, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- the University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anazodo UC, Shoemaker JK, Suskin N, St Lawrence KS. An investigation of changes in regional gray matter volume in cardiovascular disease patients, pre and post cardiovascular rehabilitation. Neuroimage Clin. 2013 Oct 6;3:388-95. doi: 10.1016/j.nicl.2013.09.011. eCollection 2013. PMID 24273722
- [Result] Barnes JN, Schmidt JE, Nicholson WT, Joyner MJ. Cyclooxygenase inhibition abolishes age-related differences in cerebral vasodilator responses to hypercapnia. J Appl Physiol (1985). 2012 Jun;112(11):1884-90. doi: 10.1152/japplphysiol.01270.2011. Epub 2012 Mar 22. PMID 22442028
- [Result] Beeri MS, Rapp M, Silverman JM, Schmeidler J, Grossman HT, Fallon JT, Purohit DP, Perl DP, Siddiqui A, Lesser G, Rosendorff C, Haroutunian V. Coronary artery disease is associated with Alzheimer disease neuropathology in APOE4 carriers. Neurology. 2006 May 9;66(9):1399-404. doi: 10.1212/01.wnl.0000210447.19748.0b. PMID 16682673
- [Result] Booth FW, Roberts CK, Laye MJ. Lack of exercise is a major cause of chronic diseases. Compr Physiol. 2012 Apr;2(2):1143-211. doi: 10.1002/cphy.c110025. PMID 23798298
- [Result] Dishman RK, Berthoud HR, Booth FW, Cotman CW, Edgerton VR, Fleshner MR, Gandevia SC, Gomez-Pinilla F, Greenwood BN, Hillman CH, Kramer AF, Levin BE, Moran TH, Russo-Neustadt AA, Salamone JD, Van Hoomissen JD, Wade CE, York DA, Zigmond MJ. Neurobiology of exercise. Obesity (Silver Spring). 2006 Mar;14(3):345-56. doi: 10.1038/oby.2006.46. PMID 16648603
- [Result] Erickson KI, Voss MW, Prakash RS, Basak C, Szabo A, Chaddock L, Kim JS, Heo S, Alves H, White SM, Wojcicki TR, Mailey E, Vieira VJ, Martin SA, Pence BD, Woods JA, McAuley E, Kramer AF. Exercise training increases size of hippocampus and improves memory. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3017-22. doi: 10.1073/pnas.1015950108. Epub 2011 Jan 31. PMID 21282661
- [Result] Filippini N, Ebmeier KP, MacIntosh BJ, Trachtenberg AJ, Frisoni GB, Wilcock GK, Beckmann CF, Smith SM, Matthews PM, Mackay CE. Differential effects of the APOE genotype on brain function across the lifespan. Neuroimage. 2011 Jan 1;54(1):602-10. doi: 10.1016/j.neuroimage.2010.08.009. Epub 2010 Aug 10. PMID 20705142
- [Result] Heli V, Ihab H, Kun H, Brad M, Jessica W, Vera N. Effects of exercise program on physiological functions in postmenopausal women with metabolic syndrome. Int J Gerontol. 2013 Dec;7(4):231-235. doi: 10.1016/j.ijge.2013.05.002. PMID 24634702
- [Result] Pires PW, Dams Ramos CM, Matin N, Dorrance AM. The effects of hypertension on the cerebral circulation. Am J Physiol Heart Circ Physiol. 2013 Jun 15;304(12):H1598-614. doi: 10.1152/ajpheart.00490.2012. Epub 2013 Apr 12. PMID 23585139
- [Result] Yates KF, Sweat V, Yau PL, Turchiano MM, Convit A. Impact of metabolic syndrome on cognition and brain: a selected review of the literature. Arterioscler Thromb Vasc Biol. 2012 Sep;32(9):2060-7. doi: 10.1161/ATVBAHA.112.252759. PMID 22895667
- [Result] Anazodo UC, Shoemaker JK, Suskin N, Ssali T, Wang DJ, St Lawrence KS. Impaired Cerebrovascular Function in Coronary Artery Disease Patients and Recovery Following Cardiac Rehabilitation. Front Aging Neurosci. 2016 Jan 5;7:224. doi: 10.3389/fnagi.2015.00224. eCollection 2015. PMID 26779011